CLINICAL TRIAL: NCT02931123
Title: A RCT COMPARING LACTULOSE AND RIFAXIMIN ASSOCIATED WITH A VEGETABLE DIET IN THE PREVENTION OF POST-TIPS OVERT HEPATIC ENCEPHALOPATHY
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof oliviero Riggio, professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OR-201
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Cirrhotic Patients Undergoing TIPS Placement
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard (No Intervention)
- treatment (Experimental): rifaximine and lattulose plus low proteine diet
  Interventions: Drug: lattulose and rifaximine

INTERVENTIONS:
Drug: lattulose and rifaximine
  Arms: treatment

SUMMARY:
This is a randomized controlled trial whose purpose is to evaluate the efficacy of therapy with lactulose and rifaximin associated with a vegetable diet in the prevention of post-TIPS hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* consecutive cirrhotic patients undergoing TIPS

Exclusion Criteria:

* age >75 years; bilirubin levels >5 mg/dl; creatinine levels >3 mg/dl; a serious cardiac or pulmonary dysfunction; a Child-Pugh's score >11 (except for the patients candidates to early TIPS); a model end-stage liver disease (MELD) score >18; a diagnosis of hepatic carcinoma; sepsis; spontaneous bacterial peritonitis; renal insufficiency. Present HE or previous spontaneous/recurrent HE, alcohol/psychoactive drugs intake (positive alcoholaemia and/or benzodiazepines or opioid urine metabolites) at the moment of evaluation, unrelated neurological disease including dementia (mini mental state < 26).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
incidence of hepatic encephalopathy | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided